CLINICAL TRIAL: NCT00926484
Title: Combined Tooth Mousse and Fluoride Varnish in Dentin Hypersensitivity Treatment
Brief Title: Tooth Mousse and Fluoride in Dentin Hypersensitivity Treatment
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Weimin Chen, Tongji Hospital, Huazhong University of Science and Technology
Other Study IDs: TF87330244
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentin hypersensitivity; Tooth Mousse; fluoride varnish
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Tooth Mousse
- fluoride varnish
- Tooth Mousse + fluoride varnish

SUMMARY:
GC Tooth Mousse, a complex containing amorphous calcium phosphate (ACP) and casein phosphopeptide (CPP), is recommended in dentin hypersensitivity reduction due to its ability to block opened dentinal tubules. It acts synergistically with fluorine in slowing caries progression. Whether CPP-ACP can act synergistically with fluorine in the dentin hypersensitivity treatment is unknown. The aim of this study was to assess the effect of CPP-ACP combined with fluoride varnish in cervical dentin hypersensitivity treatment.

ELIGIBILITY:
Inclusion Criteria:

* subjects with a minimum of three cervical hypersensitive teeth at both sides of the dental arch

Exclusion Criteria:

* dentin hypersensitivity caused by caries lesions
* fracture of restoration
* chipped teeth
* marginal gaps
* post-operative sensitivity
* cracked-tooth syndrome, and which were confirmed by periapical radiographs and teeth with cervical fillings

Ages: 26 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
ANOVA | June 2008

SECONDARY OUTCOMES:
T-test | June 2008

CONTACTS AND LOCATIONS:
Overall Officials: Xuejin Tao, Doctor, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Kowalczyk A, Botulinski B, Jaworska M, Kierklo A, Pawinska M, Dabrowska E. Evaluation of the product based on Recaldent technology in the treatment of dentin hypersensitivity. Adv Med Sci. 2006;51 Suppl 1:40-2. PMID 17458057
- See also: Treating cervical dentin hypersensitivity with fluoride varnish: a randomized clinical study. — http://www.ncbi.nlm.nih.gov/pubmed/16803829?ordinalpos=1&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum
- See also: definition of Dentine hypersensitivity — http://en.wikipedia.org/wiki/Dentine_hypersensitivity
- See also: Prevalence and distribution of cervical dentin hypersensitivity in a population in Taipei, Taiwan — http://linkinghub.elsevier.com/retrieve/pii/S0099239998802136